CLINICAL TRIAL: NCT06451588
Title: Donor Versus Autologous Fecal Microbiota Transplantation for Axial Spondyloarthritis: a Double Blind, Placebo-Controlled, Randomized Trial
Brief Title: Fecal Microbiota Transplantation in Axial Spondyloarthritis
Acronym: MicroSpA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Principal Investigator, Gunnstein Bakland, MD PhD, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 537025
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis; Dysbiosis; Spondyloarthritis; Spondylitis; Arthritis; Musculoskeletal Diseases; Spinal Disease; Joint Diseases
Keywords: Axial Spondyloarthritis; Microbiome; Fecal Microbiota Transplantation; Microbiota; FMT; RCT
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Dysbiosis; Spondylarthritis; Spondylitis; Arthritis; Musculoskeletal Diseases; Spinal Diseases; Joint Diseases

STUDY DESIGN:
Intervention Model Description: A blinded, randomized, placebo-controlled, parallel-group, single-center, superiority, phase III clinical trial. Participants randomized til active treatment will receive FMT from one of three donors. Allocation will be random in blocks of 9 (Donor A: Donor B : Donor C : Placebo 2:2:2:3).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A person will be responsible for the Randomization and Allocation (RAP) procedure, and will be the only person not blinded to randomization and treatment. This person will, however, be blinded for the patient´s identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Donor A FMT (Experimental): Active treatment contain 60g of feces from a single healthy, screened donor. The feces is combined with glycerol and saline to a total volume of 440 ml in an enema bag. Each participant will only receive a single treatment at baseline.
  Interventions: Drug: FMT
- Donor B FMT (Experimental): Active treatment contain 60g of feces from a single healthy, screened donor. The feces is combined with glycerol and saline to a total volume of 440 ml in an enema bag. Each participant will only receive a single treatment at baseline.
  Interventions: Drug: FMT
- Donor C FMT (Experimental): Active treatment contain 60g of feces from a single healthy, screened donor. The feces is combined with glycerol and saline to a total volume of 440 ml in an enema bag. Each participant will only receive a single treatment at baseline.
  Interventions: Drug: FMT
- Placebo/autologous FMT (Placebo Comparator): Placebo treatment will be processed identically to active treatment, but with paritcipants own stool. The patients in the placebo group will consequently receive an enema with 60g of their own feces combined with glycerol and saline as a single treatment at baseline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FMT — Active FMT
  Arms: Donor A FMT; Donor B FMT; Donor C FMT
Drug: Placebo — The placebo treatment will be prepared based on the patients' fecal samples (autologous).
  Arms: Placebo/autologous FMT

SUMMARY:
Although biologic therapy have revolutionized the treatment of Spondyloarthrtitis (SpA), many patients do not experience complete relief of SpA related complaints.

It has been established that patients with SpA have an altered composition of microorganisms (microbiota) in the gut compared to healthy controls, and that this correlates to disease activity and respons to therapy.

The goal of this randomized double-blind study is to evaluate the efficacy of fecal microbiota transplantation (FMT) in patients with axial SpA with a suboptimal effect of biologic therapy.

The main questions it aims to answer are:

* Can FMT reduce disease activity in axial SpA?
* Can FMT alleviate pain and reduce fatigue in axial SpA?
* Is the composition of microorganisms restored to normal in patients with SpA after a treatment with FMT?

Participants will receive a single treatment in the form of an enema with either donor FMT or placebo at baseline. The primary endpoint will be evaluated after 90 days, but efficacy and safety will be monitored from baseline until 365 days.

DETAILED DESCRIPTION:
Axial Spondyloarthritis (axSpA) is a chronic inflammatory disease affecting the sacroiliac joints (SIJ) and the spine.

The approach to treatment of axSpA is a combination of patient education, with a focus on exercise and lifestyle, and a medical treatment. Non-steroidal anti-inflammatory drugs (NSAIDs) are the first-line medical treatment, providing symptom relief for a large portion of the patients. For patients with inadequate response, or intolerance, to NSAIDs, biological (TNFi and IL17i) or targeted synthetic (JAKi) disease modifying drugs (b/ts-DMARDs) are considered a second-line treatment option and provide excellent efficacy for many patients. However, a substantial portion of the patients experience active disease despite this second-line therapy.

The cause of the disease is multifactorial, and both genetic and environmental factors contribute in the pathogenesis. Patients with axSpA have a higher prevalence of inflammatory bowel disease (IBD) than the background population, i.e. Crohn's disease and ulcerative colitis. However, inflammation in the gut is also demonstrated in 50-70% of patients without symptoms of IBD, and this inflammation is believed to be of importance in the development of the disease.

The human gut microbiota is the collection of microbes in the intestines. The composition of the microbiota is the result of many factors and have evolved over time to form a mutually beneficial relationship to both humans and microorganisms. Normally there is a balance and a stability in this composition, but in many conditions an imbalance, termed dysbiosis, has been demonstrated. This is also the case in axSpA, and the extent of this dysbiosis also relates to disease activity and to response to therapy.

Fecal microbiota transplantation (FMT) is a method used to alter the microbiota composition by transferring microbes from a healthy individual to a recipient. In several conditions this has both proven the ability to alter the microbiota and to provide symptom relief , e.g. clostridium difficile infections, ulcerative colitis and irritable bowel syndrome.

Given the potential role of the microbiota in the pathogenesis of axSpA, we wish to evaluate whether replacing the microbiota in patients with inadequate response to biologic therapy with FMT can be efficacious in providing a state of inactive disease and symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* Axial Spondyloarthritis according to the ASAS classification criteria
* Active disease defined as ASDAS ≥2.1 with elevated CRP ≥4 OR active inflammation on MRI within the last 3 months
* Onset of axial SpA within last 10 years
* Unsatisfactory relief of NSAIDs
* On stable immunomodulatory treatment (TNFi, IL17i or JAKi) the last 3 months

Exclusion Criteria:

* Planned dose adjustment or change in immunomodulatory treatment the next 90 days
* Disease or disorder with life expectancy of ≤5 years
* Severe immune deficiency (acquired, congenital og du to medication)
* Previous treatment with FMT
* Regular use of opioids with the exception of codeine and tramadol
* Any specific diagnosis that could explain or contribute to the patients back pain (e.g. tumor, fracture, infection or degenerative disease)
* Inflammatory spinal disease other than axSpA
* Severe psychiatric disorder, alcohol- or drug abuse
* Active inflammatory bowel disease
* Microscopic colitis, diverticulitis or ileus
* Active psoriasis
* Fibromyalgia
* Abdominal surgery excluding appendectomy, cholecystectomy, hysterectomy, caesarian section, sapling-ooforectomy and hernia surgery
* Malignant disease excluding basalioma and melanoma stage 1
* Conditions with expected necessary treatment with antibiotics during the study period, e.g. periodontitis end ischemic digital ulcers
* Treatment with antibiotics 12 weeks prior to study entry
* Pregnancy, lactation or planned pregnancy within the next 3 months
* Contraindications for rectal catheter insertion
* Planned rehabilitation program the next 90 days
* Limited ability to comply with protocol requirements, including biobank participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Minimal Clinically Important Improvement | 90 days
  Proportion of patients that meet the criteria of Minimal Clinically Important Improvement in the donor FMT (dFMT) versus the autologous FMT (aFMT) group at day 90 after treatment. Minimal Clinically Important Improvement is defined by a decrease of ≥1,1 in ASDAS-CRP

SECONDARY OUTCOMES:
Adverse events | Day 0-90 and day 91-365
  The proportion of patients experiencing any adverse events from baseline util day 90 and day 365
Ankylosing Spondylitis Disease Activity Score (ASDAS)20 | baseline, day 30, day 60 and day 90
  Change in the dFMT vs aFMT group from baseline
Bath Ankylosing Spondylitis Disease Activity Index | baseline, day 30, day 60 and day 90
  Change in the dFMT vs aFMT group from baseline
Bath Anykylosing Spondylitis Funtional Index | baseline, day 30, day 60 and day 90
  Change in the dFMT vs aFMT group from baseline
Patient global assessment | baseline, day 30, day 60 and day 90
  Change in the dFMT vs aFMT group from baseline
VAS spinal pain | baseline, day 30, day 60 and day 90
  Change in the dFMT vs aFMT group from baseline
Modified Fatigue Impact Scale | baseline and day 90
  Change in the dFMT vs aFMT group from baseline
RAND-36 | baseline and day 90
  Change in the dFMT vs aFMT group from baseline
Maastricht Ankylosing Spondylitis Enthesitis Score | baseline and day 90
  Change in the dFMT vs aFMT group from baseline
The 66/68 Joint Count Score | baseline and day 90
  Change in the dFMT vs aFMT group from baseline
Bath Ankylosing Spondylitis Metrology Index | baseline and day 90
  Change in the dFMT vs aFMT group from baseline
Ankylosing Spondylitis Disease Activity Score (ASDAS)40 | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
Bath Ankylosing Spondylitis Disease Activity Index | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
Bath Anykylosing Spondylitis Funtional Index | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
Patient global assessment | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
VAS spinal pain | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
Modified Fatigue Impact Scale | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline
RAND-36 | baseline and day 30, day 60, day 90, day 180, day 270 and day 365
  Long term change that includes the extended open labeled follow up in the dFMT vs aFMT group from baseline

OTHER OUTCOMES:
Exploratory endpoint | baseline and day 90
  Changes in taxonomy and function of the microbiome, the immune system, metabolome and gut epithelial barrier in participants with vs without treatment success to dFMT and aFMT
Exploratory endpoint | baseline
  Differences in baseline taxonomy and function of the microbiome, the immune system, metabolome and gut epithelial barrier in participants with vs without treatment success to dFMT and aFMT

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
There is not an IPD established.

REFERENCES:
- [Result] Baraliakos X, Braun J. Spondyloarthritides. Best Pract Res Clin Rheumatol. 2011 Dec;25(6):825-42. doi: 10.1016/j.berh.2011.11.006. PMID 22265264
- [Result] Zheng D, Liwinski T, Elinav E. Interaction between microbiota and immunity in health and disease. Cell Res. 2020 Jun;30(6):492-506. doi: 10.1038/s41422-020-0332-7. Epub 2020 May 20. PMID 32433595
- [Result] Imdad A, Nicholson MR, Tanner-Smith EE, Zackular JP, Gomez-Duarte OG, Beaulieu DB, Acra S. Fecal transplantation for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2018 Nov 13;11(11):CD012774. doi: 10.1002/14651858.CD012774.pub2. PMID 30480772
- [Result] Bazin T, Hooks KB, Barnetche T, Truchetet ME, Enaud R, Richez C, Dougados M, Hubert C, Barre A, Nikolski M, Schaeverbeke T. Microbiota Composition May Predict Anti-Tnf Alpha Response in Spondyloarthritis Patients: an Exploratory Study. Sci Rep. 2018 Apr 3;8(1):5446. doi: 10.1038/s41598-018-23571-4. PMID 29615661
- [Result] Johnsen PH, Hilpusch F, Cavanagh JP, Leikanger IS, Kolstad C, Valle PC, Goll R. Faecal microbiota transplantation versus placebo for moderate-to-severe irritable bowel syndrome: a double-blind, randomised, placebo-controlled, parallel-group, single-centre trial. Lancet Gastroenterol Hepatol. 2018 Jan;3(1):17-24. doi: 10.1016/S2468-1253(17)30338-2. Epub 2017 Nov 1. PMID 29100842
- [Result] Breban M, Beaufrere M, Glatigny S. The microbiome in spondyloarthritis. Best Pract Res Clin Rheumatol. 2019 Dec;33(6):101495. doi: 10.1016/j.berh.2020.101495. Epub 2020 Mar 12. PMID 32173258